CLINICAL TRIAL: NCT00099164
Title: A Randomized Trial of 17 Alpha-Hydroxyprogesterone Caproate for Prevention of Preterm Birth in Multifetal Gestation (STTARS)
Brief Title: Trial of Progesterone in Twins and Triplets to Prevent Preterm Birth (STTARS)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: The George Washington University Biostatistics Center (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: HD36801-STTARS; HD21410; HD27869; HD27917; HD27860; HD27915; HD34116; HD34208; HD34136; HD40500; HD40485; HD40544; HD40545; HD40560; HD40512; HD36801
Record Dates: First submitted 2004-12-08; First posted 2004-12-09 (Estimated); Last update posted 2019-02-21 (Actual); Status verified 2019-02

CONDITIONS: Preterm Birth; Pregnancy; Multifetal
Keywords: preterm birth; pregnancy; multifetal; Progesterone
MeSH Terms: conditions — Premature Birth | interventions — 17 alpha-Hydroxyprogesterone Caproate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: 17 alpha-hydroxyprogesterone caproate (17P) — Study coded medication is 250 mg of 17P as a 1 ml intramuscular injection (or 1 ml of placebo inert oil). Patients are seen weekly to administer the study drug through 34 weeks 6 days gestation or delivery, whichever occurs first.

SUMMARY:
Women pregnant with twins or triplets are at high risk of preterm birth, yet no intervention or approach has served to reduce this risk. A recently completed trial by the NICHD sponsored Maternal Fetal Medicine Units (MFMU) Network has, for the first time, demonstrated a treatment that substantially reduces the rate of preterm birth in women at high risk for preterm delivery (i.e. progesterone therapy). Preterm birth was reduced by 35% among progesterone-treated women with a singleton pregnancy when compared with women receiving placebo. The current trial compares weekly treatment by injection of progesterone with placebo in women pregnant with twins or triplets.

DETAILED DESCRIPTION:
Women with multifetal gestation face numerous risks in excess of those faced by women with singleton gestation. Preterm birth is by far the most common and the most significant of these problems, yet no intervention or approach has served to reduce this risk. The prevalence of preterm birth has risen dramatically in recent years, in large part due to Assisted Reproductive Technologies. Consequently, the problem of preterm birth has assumed an even greater role in contributing to perinatal morbidity and mortality. The recently completed trial by the NICHD sponsored Maternal Fetal Medicine Units (MFMU) Network has, for the first time, demonstrated a treatment (i.e. progesterone therapy) that substantially reduces the rate of preterm birth in women at high risk for preterm delivery because of a prior spontaneous preterm birth . Preterm birth was reduced by 35% among progesterone-treated women when compared with women receiving placebo. Given this dramatic benefit and the extremely high risk of preterm birth in women with multifetal gestation, a trial to evaluate the benefit of progesterone in women with multifetal pregnancy is appropriate and timely. This protocol outlines a randomized, double-masked clinical trial comparing weekly treatment by injection of 17 alpha-hydroxyprogesterone caproate (17P) with placebo in women with twin or triplet gestation. In an ancillary study, the pharmacokinetics and pharmacodynamics of 17P in multifetal gestation will be studied.

This trial aims to enroll six hundred women with twin gestation and one hundred twenty women with triplet gestation between 16 weeks 0 days to 20 weeks 6 days. At the initial screening evaluation, and after signing the informed consent form, the patient will receive an injection of the placebo (1 ml inert castor oil). She will be asked to return after three days for randomization. During this compliance test period, an ultrasound exam will be scheduled, if not previously done. When the patient returns and if she still meets the inclusion criteria, she will be randomized to one of two treatments:

* 17 a-hydroxyprogesterone caproate: weekly 1 ml injections containing 250 mg of 17P
* Placebo: weekly injections of 1 ml placebo inert castor oil

Treatment will be given through 34 weeks 6 days gestation or delivery. At the time of consent to the main study, the patient will also be asked to participate in an ancillary study. If she agrees, she will have 30 cc of blood drawn at 24-28 weeks and at 32-35 weeks gestation. A pelvic exam will be done at the same two times to collect vaginal specimens and to determine Bishop score.

ELIGIBILITY:
Inclusion Criteria:

* Twin or triplet pregnancy. Quadruplets reduced to triplets may be included, but no other prior reductions.
* Gestational age between 16 weeks 0 days to 20 weeks 6 days based on clinical information and evaluation of the first ultrasound.
* Signed patient authorization and consent form.

Exclusion Criteria:

* Prior elective fetal reduction in the current pregnancy, except in the case of a quadruplet gestation reduced to triplets.
* Planned fetal reduction or planned termination
* Monoamniotic gestation
* Twin-twin transfusion syndrome
* Fetal death or imminent fetal demise
* Major fetal anomaly (e.g., gastroschisis, spina bifida, serious karyotypic abnormalities). An ultrasound examination from 12 weeks 0 days to 20 weeks 6 days by project estimated date of confinement (EDC) must be performed to rule out fetal anomalies
* Discordance in fetal size, defined as a discrepancy of 3 or more weeks in gestational age by ultrasound between the largest and the smallest fetus. Diagnosis is based on measurements made at the ultrasound done between 12 weeks 0 days and 20 weeks 6 days gestation
* Progesterone treatment used or planned after 14 weeks gestation
* Heparin therapy at a dose ≥ 10,000 units per day of unfractionated heparin, or any low molecular weight heparin during the current pregnancy, or thromboembolic disease for which such heparin treatment is planned (because of contraindication to intra-muscular injections)
* Current or planned cervical cerclage
* Uterine anomaly (uterine didelphys, bicornate uterus)
* Contraindication to intra-muscular injections
* Maternal medical conditions, such as: known idiopathic thrombocytopenia purpura (ITP) or a known platelet count less than 100,000 per cubic millimeter (because of contraindication to intra-muscular injections), hypertension requiring medication, diabetes managed with insulin or oral hypoglycemic agents
* Inability to arrange a pre-randomization ultrasound between 12 weeks 0 days and 20 weeks 6 days gestation
* Participation in another interventional study that influences gestational age at delivery or neonatal morbidity or mortality
* Prenatal follow-up or delivery planned elsewhere (unless the study visits can be made as scheduled and complete outcome information can be obtained)
* Participation in this trial in a previous pregnancy.

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 795 (Actual)
Dates: Start 2004-04; Primary Completion 2006-08 (Actual); Study Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
Delivery prior to 35 weeks 0 days gestation | Delivery Date

SECONDARY OUTCOMES:
Maternal randomization to delivery interval of first fetus | Delivery
pPROM - spontaneous rupture of the membranes at least one hour prior to the start of labor, regular contractions accompanied by cervical change | Duration of pregnancy
Indicated preterm delivery | Delivery
Spontaneous preterm delivery | Delivery
Cesarean delivery | Delivery
Gestational age at delivery | Length of pregnancy
Placement of cervical cerclage | During pregnancy
Maternal hospital days | Delivery
Maternal complications such as preeclampsia, gestational diabetes, placental abruption, chorioamnionitis. | Duration of pregnancy, delivery
Composite neonatal outcome, comprised of fetal or infant death, RDS, IVH (grades 3 and 4), PVL, NEC (stage II and III), BPD/chronic lung disease, ROP (stage III or higher), early onset sepsis including meningitis | Early life
Fetal and neonatal death | Delivery, Early life
Stillbirth | Delivery
Twin-twin transfusion syndrome | During pregnancy
Birth weight and degree of birth weight discordance | Birth
Infant days in hospital, *Respiratory distress syndrome (RDS) | Early life
Transient tachypnea of the newborn (TTN) | Early life
Bronchopulmonary dysplasia (BPD)/chronic lung disease | Early life
Persistent pulmonary hypertension of the newborn (PPHN) | Early life
Duration of ventilator support | Early life
Duration of supplemental oxygen | Early life
Periventricular leukomalacia (PVL) | Early life
Intraventricular hemorrhage (IVH) | Early life
Necrotizing enterocolitis (NEC) | Early life
Neonatal sepsis/meningitis/urinary tract infection/ pneumonia | Early life
Seizures, as documented by the attending physician | Early life
Retinopathy of prematurity (ROP) | Early life
Small for gestational age (<10th percentile). | Early life

CONTACTS AND LOCATIONS:
Overall Officials: Menachem Miodovnik, M.D., Study Director — NICHD Project Scientist; Elizabeth A Thom, Ph.D., Principal Investigator — George Washington University Biostatistics Center; Dwight Rouse, MD, Study Chair — University of Alabama at Birmingham; Steve N Caritis, MD, Study Chair — University of Pittsburgh - Magee Womens Hospital
Locations (14):
- United States (14):
  - University of Alabama - Birmingham, Birmingham, Alabama
  - Northwestern University, Chicago, Illinois
  - Wayne State University, Detroit, Michigan
  - Columbia University, New York, New York
  - University of North Carolina - Chapel Hill, Chapel Hill, North Carolina
  - Wake Forest University School of Medicine, Winston-Salem, North Carolina
  - Case Western University, Cleveland, Ohio
  - Ohio State University, Columbus, Ohio
  - Dexel University, Philadelphia, Pennsylvania
  - University of Pittsburgh Magee Womens Hospital, Pittsburgh, Pennsylvania
  - Brown University, Providence, Rhode Island
  - University of Texas - Southwest, Dallas, Texas
  - University of Texas - Houston, Houston, Texas
  - University of Utah Medical Center, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: Yes
The data will be shared after completion and publication of the main analyses in accordance with NIH policy. The dataset can be obtained by emailing mfmudatasets@bsc.gwu.edu.

REFERENCES:
- [Background] Meis PJ, Klebanoff M, Thom E, Dombrowski MP, Sibai B, Moawad AH, Spong CY, Hauth JC, Miodovnik M, Varner MW, Leveno KJ, Caritis SN, Iams JD, Wapner RJ, Conway D, O'Sullivan MJ, Carpenter M, Mercer B, Ramin SM, Thorp JM, Peaceman AM, Gabbe S; National Institute of Child Health and Human Development Maternal-Fetal Medicine Units Network. Prevention of recurrent preterm delivery by 17 alpha-hydroxyprogesterone caproate. N Engl J Med. 2003 Jun 12;348(24):2379-85. doi: 10.1056/NEJMoa035140. PMID 12802023
- [Background] Kogan MD, Alexander GR, Kotelchuck M, MacDorman MF, Buekens P, Papiernik E. A comparison of risk factors for twin preterm birth in the United States between 1981-82 and 1996-97. Matern Child Health J. 2002 Mar;6(1):29-35. doi: 10.1023/a:1014312132443. PMID 11926251
- [Background] Gardner MO, Goldenberg RL, Cliver SP, Tucker JM, Nelson KG, Copper RL. The origin and outcome of preterm twin pregnancies. Obstet Gynecol. 1995 Apr;85(4):553-7. doi: 10.1016/0029-7844(94)00455-M. PMID 7898832
- [Background] Min SJ, Luke B, Gillespie B, Min L, Newman RB, Mauldin JG, Witter FR, Salman FA, O'sullivan MJ. Birth weight references for twins. Am J Obstet Gynecol. 2000 May;182(5):1250-7. doi: 10.1067/mob.2000.104923. PMID 10819867
- [Background] Lynch A, McDuffie R, Stephens J, Murphy J, Faber K, Orleans M. The contribution of assisted conception, chorionicity and other risk factors to very low birthweight in a twin cohort. BJOG. 2003 Apr;110(4):405-10. PMID 12699803
- [Background] Goldenberg RL, Iams JD, Miodovnik M, Van Dorsten JP, Thurnau G, Bottoms S, Mercer BM, Meis PJ, Moawad AH, Das A, Caritis SN, McNellis D. The preterm prediction study: risk factors in twin gestations. National Institute of Child Health and Human Development Maternal-Fetal Medicine Units Network. Am J Obstet Gynecol. 1996 Oct;175(4 Pt 1):1047-53. doi: 10.1016/s0002-9378(96)80051-2. PMID 8885774
- [Result] Caritis SN, Rouse DJ, Peaceman AM, Sciscione A, Momirova V, Spong CY, Iams JD, Wapner RJ, Varner M, Carpenter M, Lo J, Thorp J, Mercer BM, Sorokin Y, Harper M, Ramin S, Anderson G; Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD), Maternal-Fetal Medicine Units Network (MFMU). Prevention of preterm birth in triplets using 17 alpha-hydroxyprogesterone caproate: a randomized controlled trial. Obstet Gynecol. 2009 Feb;113(2 Pt 1):285-92. doi: 10.1097/AOG.0b013e318193c677. PMID 19155896
- [Result] Rouse DJ, Caritis SN, Peaceman AM, Sciscione A, Thom EA, Spong CY, Varner M, Malone F, Iams JD, Mercer BM, Thorp J, Sorokin Y, Carpenter M, Lo J, Ramin S, Harper M, Anderson G; National Institute of Child Health and Human Development Maternal-Fetal Medicine Units Network. A trial of 17 alpha-hydroxyprogesterone caproate to prevent prematurity in twins. N Engl J Med. 2007 Aug 2;357(5):454-61. doi: 10.1056/NEJMoa070641. PMID 17671253
- [Result] Gyamfi C, Horton AL, Momirova V, Rouse DJ, Caritis SN, Peaceman AM, Sciscione A, Meis PJ, Spong CY, Dombrowski M, Sibai B, Varner MW, Iams JD, Mercer BM, Carpenter MW, Lo J, Ramin SM, O'Sullivan MJ, Miodovnik M, Conway D; Eunice Kennedy Shriver National Institute of Child Health and Human Development Maternal-Fetal Medicine Units Network. The effect of 17-alpha hydroxyprogesterone caproate on the risk of gestational diabetes in singleton or twin pregnancies. Am J Obstet Gynecol. 2009 Oct;201(4):392.e1-5. doi: 10.1016/j.ajog.2009.06.036. Epub 2009 Aug 29. PMID 19716543
- [Derived] Blumenfeld YJ, Momirova V, Rouse DJ, Caritis SN, Sciscione A, Peaceman AM, Reddy UM, Varner MW, Malone FD, Iams JD, Mercer BM, Thorp JM Jr, Sorokin Y, Carpenter MW, Lo J, Ramin SM, Harper M; Eunice Kennedy Shriver National Institute of Child Health and Human Development Maternal-Fetal Medicine Units Network. Accuracy of sonographic chorionicity classification in twin gestations. J Ultrasound Med. 2014 Dec;33(12):2187-92. doi: 10.7863/ultra.33.12.2187. PMID 25425377
- [Derived] Caritis SN, Sharma S, Venkataramanan R, Rouse DJ, Peaceman AM, Sciscione A, Spong CY, Varner MW, Malone FD, Iams JD, Mercer BM, Thorp JM Jr, Sorokin Y, Carpenter M, Lo J, Ramin S, Harper M; Eunice Kennedy Shriver National Institute of Child Health and Human Development Maternal-Fetal Medicine Units Network. Pharmacokinetics of 17-hydroxyprogesterone caproate in multifetal gestation. Am J Obstet Gynecol. 2011 Jul;205(1):40.e1-8. doi: 10.1016/j.ajog.2011.03.028. Epub 2011 Mar 22. PMID 21620357
- See also: The public website of the NICHD Maternal Fetal Medicine Units (MFMU) Network — http://www.bsc.gwu.edu/mfmu/